CLINICAL TRIAL: NCT01510977
Title: The Outcome of a Second Preparation for Colonoscopy After Preparation Failure in the First Procedure: a Prospective Randomized Controlled Study
Brief Title: Second Bowel Preparation for Colonoscopy Failure
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jeong-Sik Byeon, Clinical Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2009-0733
Record Dates: First submitted 2012-01-09; First posted 2012-01-18 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Colonoscopy Failure; Poor Bowel Preparation
Keywords: colonoscopy; bowel preparation
MeSH Terms: interventions — Polyethylene Glycols; Bisacodyl

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEG (Active Comparator): 2L of polyethylene glycol addition immediately after first colonoscopy failure
  Interventions: Drug: polyethylene glycol
- PEG + bisacodyl (Experimental): One week after initial colonoscopy failure, conventional amount (5L) of polyethylene glycol together with bisacodyl administration
  Interventions: Drug: polyethylene glycol, Bisacodyl

INTERVENTIONS:
Drug: polyethylene glycol, Bisacodyl — After failure of first colonoscopy, bowel preparation with polyethylene glycol and bisacodyl one week after
  Arms: PEG + bisacodyl
Drug: polyethylene glycol — Immediately after first colonoscopy failure, polyethylene glycol 2L addition
  Arms: PEG

SUMMARY:
Colonoscopy is a basic but important tool to diagnose and treat lesions of the colon. Proper colon cleansing is essential for colonoscopy to be performed with a good quality. Inadequate bowel preparation leads to longer colonoscopic insertion time and patient discomfort, as well as inadequate diagnostic yield of colonic lesions. Frequency of colonoscopy failure due to bad bowel preparation is reported to be 0.3% to 6.5 percent, and the rate increases with liver cirrhosis, constipation, dementia, stroke, or administration of tricyclic antidepressants. In case of colonoscopy failure due to bad bowel preparation, the second colonoscopy can be performed with either adding a colon cleansing solution immediately, or it can be performed after a few days with colon cleansing agent together with prokinetics. These different kinds of bowel preparations after first colonoscopy failure have not been compared.

ELIGIBILITY:
Inclusion Criteria:

* First colonoscopy failure due to inadequate bowel preparation

Exclusion Criteria:

* younger than 18 years old
* presence of inflammatory bowel disease
* pregnant
* lactating
* refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
second colonoscopy failure due to inadequate bowel preparation (PEG+bisdacodyl group) | one week
second colonoscopy failure due to inadequate bowel preparation (PEG group) | within the same day

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Sik Byeon, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea